CLINICAL TRIAL: NCT00484835
Title: Randomised Control Trial Comparing Hysterectomy Using Electrocoagulation Forceps With the Traditional Clamp & Suture Technique of Richardson Abdominal Hysterectomy
Brief Title: Are Sutures Required in Total Abdominal Hysterectomy? A Randomised Control Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southern Health (Other)
Collaborators: Gyrus ACMI (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Electrocoag Forceps in TAH
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-06

CONDITIONS: Total Abdominal Hysterectomy
Keywords: Abdominal; Hysterectomy; Electrocoagulation forceps; Electrosurgery; Gyrus plasma open seal forceps; Patients undergoing abdominal hysterectomy for various reasons
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Performing abdominal hysterectomy using gyrus electrocoagulation forceps

SUMMARY:
The Hypothesis of this study is that performing total abdominal hysterectomy using the newer electrocoagulation forceps, specifically, the gyrus open seal forceps, curved, compared to the traditional clamp & suture technique will result in reduction of operating time, intra-operative blood loss, post-operative pain.

DETAILED DESCRIPTION:
Patients booked for total abdominal hysterectomy in Southern Health will be offered participation in the trial, and randomised to two groups: one group undergoing the procedure with the gyrus forceps & the other group with the traditional clamp & suture method. Each patient will receive detailed information regarding the study both in document form as well as verbally by the Gynaecology doctors in the pre-admission clinic prior to obtaining consent.

The researcher will collect relevant data including age of patient, medical & surgical history and data relating to both the primary & secondary outcome measures, which include length of operation, intra-operative blood loss,post-operative pain measures as well as length of hospital stay & cost.

A qualified statistician will perform power calculations and analyse the data collected, looking at the outcome measures mentioned above.

Electrical surgery has been used extensively in surgery, especially in laparoscopic surgery, and the use of these newer electrocoagulation forceps that can simultaneously haemostatically seal & cut tissue is again well established in laparoscopic surgery but only more recently introduced to open surgical procedures. To date, except for 1 pilot study, there are no randomised control trials that confirm the proposed benefits of these newer device in abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient already on waitlist in Southern Health for abdominal hysterectomy with suspected benign pathology

Exclusion Criteria:

* Patients without consent and/or with suspected malignant pathology

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Operating time, Blood loss, Post-operative pain | 1 year

SECONDARY OUTCOMES:
Length of hospital stay, Cost of the procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marziya Kadir, MBBS, Principal Investigator — Southern Health
Locations (3):
- Australia (3):
  - Casey Hospital, Melbourne, Victoria
  - Dandenong Hospital, Melbourne, Victoria
  - Monash Medical Centre(Moorabin), Melbourne, Victoria